CLINICAL TRIAL: NCT03221647
Title: A Gliadin Peptide Regulated the INF-α Immune Response in Celiac Small Intestine and in an En-terocyte Cell Line
Brief Title: INF-α Innate Immune Response to Gliadin
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, M. Vittoria Barone, Professor, Federico II University
Other Study IDs: Innate immunity CD
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; P31-43; Loxorubine; TLR7.
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Intestinal biopsies from CD patients and controls obtained during routine analysis. Informed consensus statement obtained from all subjects or their tutors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: Intestinal biopsies from controls, affected by gastroesophageal reflux,
  Interventions: Other: Intestinal biopsies
- GCD CD (Gluten Containing Diet CD): Intestinal biopsies from GFD patients had with negative serology (anti-tTg antibodies between 0 and 1.5 U/ml and EMA negative) and normal biopsy (Marsh T0-1).
  Interventions: Other: Intestinal biopsies
- GFD CD (Gluten Free Diet CD): Intestinal biopsies from GCD-CD patients with villous atrophy (Marsh T3a-c) had positive serology (anti-tTg antibodies >30 U/ml and EMA positive) ).
  Interventions: Other: Intestinal biopsies

INTERVENTIONS:
Other: Intestinal biopsies — Intestinal biopsies obtained from Patients and Controls by EGDS. The patients and controls had the intestinal biopsies as a diagnostic step or routine check independently from the present study. For this study 3 additional biopsies samples were done in patients and controls that signed the informed consent.

SUMMARY:
Background & Aims The enteropathy in Celiac Disease (CD) is due the adaptive and to the innate immune response to gliadin peptides. Gliadin peptide P31-43 activates innate immune response and interferes with vesicular trafficking. Type 1 interferons (INFs) and viral infections play a role in CD pathogenesis. In this paper investigators investigated the role of P31-43 in the activation of the INF-α pathway.

Methods Small intestinal biopsies of CD patients both with active disease on gluten containing diet (GCD) and in remission phase of the disease on a gluten free diet (GFD) and controls were analyzed before and after culture with P31-43. The levels of toll like receptor 7 (TLR7), myeloid differentiation primary response 88 (MyD88), myxovirus resistance protein 1 (MxA) and nuclear factor-κB (NF-κB) proteins and INF-α mRNA was analyzed in intestinal biopsies.

DETAILED DESCRIPTION:
Intestinal biopsies from CD patients and controls were obtained after EGDS performed during routine analysis. The biopsies were immediately immersed in culture medium (Dulbecco's modified medium, DMEM) in a falcon tube and kept for 16h at 37 C before cultivation. Biopsies were cultivated as described in Barone MV1, Caputo I, Ribecco MT, Maglio M, Marzari R, Sblattero D, Troncone R, Auricchio S, Esposito C. Humoral immune response to tissue transglutaminase is related to epithelial cell proliferation in celiac disease. Gastroenterology. 2007,132(4):1245-53.

ELIGIBILITY:
Inclusion Criteria:

biopsy fragments from duodenum were obtained from CD patients with villous atrophy on GCD, controls, affected by gastroesophageal reflux, and CD patients on GFD.

Exclusion Criteria:

other inflammatory intestinal diseases

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: For organ culture studies, biopsy fragments from duodenum were obtained from CD patients with villous atrophy on GCD, controls, affected by gastroesophageal reflux, and CD patients on GFD. Age range for all subjects was 2-17 years.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Mxa and INF alpha proteins in CD biopsies compared to controls | through study completion, an average of 1 year
  Intestinal biopsies from CD patients and controls were used to study protein levels of MxA and INF-alpha by western blot. MxA protein levels were compared to tubulin and ERK as loading control. Student t test was used to analyse the data.

CONTACTS AND LOCATIONS:
Overall Officials: M.Vittoria Barone, Principal Investigator — Federico II University
Locations (1):
- Riccardo Troncone, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
The statistical data concerning the intestinal biopsies will be published on international journal
Time Frame: the statistical analysis will be published
Access Criteria: Publication on international journal